CLINICAL TRIAL: NCT02898285
Title: Promoting Sport Participation During Early Parenthood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Victoria (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Primary Investigator, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BC16-207
Record Dates: First submitted 2016-08-30; First posted 2016-09-13 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Parents; Well-being

ARMS (3):
- Personal time condition (Active Comparator): People randomized to this group will be asked to go on a "night out" with no kids (i.e. dinner, or a movie) once a month.
  Interventions: Behavioral: Night out
- Individual sport condition (Experimental): People randomized to this group will select an individual sport. They will be asked to participate in this individual sport for three months.
  Interventions: Behavioral: Individual sport condition
- Team sport condition (Experimental): People randomized to this group will select a team sport. They will be asked to participate in the team sport for three months (length of the team sport season).
  Interventions: Behavioral: Team sports

INTERVENTIONS:
Behavioral: Team sports — Participants will choose from a list of team sports and will be signed up with the team.
  Arms: Team sport condition
Behavioral: Individual sport condition — Participants will choose from a list of individual sports.
  Arms: Individual sport condition
Behavioral: Night out — Participants in this group will be asked to go out to have a weekly night out or "personal time" of choice, such as dinner or a movie (only restrictions are they cannot go do a sport or physical activity and time must be spent without children).
  Arms: Personal time condition

SUMMARY:
The primary objective of this investigation is to test the efficacy of two sport participation formats (individual sport, team sport) on key psychosocial outcomes compared to a non-sport condition among parents of young children who were not participating in sport at baseline of the study.

Research of this type is important because parents represent a group dealing with numerous challenges and this is a period of time shown to have the greatest decline in physical activity. Furthermore, parents could reap great benefits in psychological health through the increase in physical activity and sport participation.

It is hypothesized that participation will be predicted by sports commitment as per the tenets of the Sport Commitment Model, and commitment will be predicted primarily by enjoyment (+), social constraints from family obligations/involvement alternatives (-), followed by social involvement opportunities/personal investments (+).

DETAILED DESCRIPTION:
This study is exploring the impact team sports has on psychological well-being of parents compared to individual sports or "personal time". Our research questions include:

Does 1) team sports participation (choice-based from existing adult recreation leagues in greater Victoria) increase psychosocial outcomes (quality of life, relationship satisfaction, social functioning, perceived parenting capability, enjoyment) compared with 2) individual sport participation (choice-based from adult recreation alternatives in greater Victoria), and 3) a control condition? Hypothesis: The team sports condition will show significantly larger changes in psychosocial outcomes compared to the two other conditions after three-months of participation (primary end-point). Furthermore, the individual sports condition will show significantly larger changes in psychosocial outcomes compared to the control condition after three-months of participation.

Secondary Research Questions

1. Can participation in the team sports and individual sports conditions be explained by the constructs of the Sport Commitment model [21]? Hypothesis: Participation will be predicted by sports commitment as per the tenets of the Sport Commitment Model, and commitment will be predicted primarily by enjoyment (+), social constraints from family obligations/involvement alternatives (-), followed by social involvement opportunities/personal investments (+).
2. Can group differences among parents with regard to these participation and psychosocial outcomes be explained through a mediation model? Hypothesis: The covariance of the assigned conditions on psychosocial outcomes will be explained by sport participation. In turn, the covariance between participation and assigned conditions will be explained by salient underlying motives from the Sport Commitment Model. In particular, enjoyment will explain the differences between both sport conditions but the better psychosocial outcomes from team sports will be explained by the additional social involvement opportunities.
3. Is there a seasonal, gender, dual/single parent, age of child, or type of sport difference across primary outcomes by assigned condition? Hypothesis: These are exploratory research questions with no pre-set hypothesis. Both sport conditions may have participation lowered by weather conditions in the winter. Men may participate in sport more due to lower child-rearing expectations but there is limited research to support this conjecture at this time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with children under the age of 13 who live in the Greater Victoria area
* Must not have participated in any organized sport within the last month

Exclusion Criteria:

* Parents who do not have a child under the age of 13
* Parents who have or are currently playing an organized sport
* Parents under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-10; Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in Parental Quality of Life | Baseline, six weeks and three months
  Short Form 12 Health Survey will be administered in the baseline questionnaire
Change in life satisfaction | Baseline, six weeks, and three months
  Satisfaction with Life Scale will be examined at baseline. Citation: Diener E., Emmons R. A., Larsen R. J., Griffin S. (1985). The satisfaction with life scale. Journal of Personality Assessment, 49, 71-75.
Change in Parenting Stress | Baseline, six weeks and three months
  Berry, JD, & Jones, W,H, (1995) The Parental Stress Scale : initial psychometric evidence. Journal of Social and Personal Relationships, 12, 463 - 472.

SECONDARY OUTCOMES:
Sport Commitment Model Questionnaire (Scanlan, 1993) | baseline, six-weeks, three months
  Questionnaire measure from Scanlan, 1993
Family functioning questionnaire | baseline, six weeks, three months
  35 item questionnaire from Beavers, W. R., & Hampson, R. B. (1990). Successful families: Assessment and intervention. New York: Norton.
Relationship Satisfaction questionnaire | baseline, six weeks, three months
  Relationship Assessment Scale Hendrick, S. S., Dicke, A., & Hendrick, C. (1998). The relationship assessment scale. Journal of Social and Personal Relationships, 15(1), 137-142.
  HarperCollins.

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioural Medicine Laboratory, Victoria, British Columbia, Canada

REFERENCES:
- [Derived] Rhodes RE, Beauchamp MR, Carson V, Courtnall S, Wierts CM, Blanchard CM. Effect of recreational sport and physical activity participation on well-being during early parenthood: a randomized controlled trial. Ann Behav Med. 2025 Jan 4;59(1):kaae081. doi: 10.1093/abm/kaae081. PMID 39657760
- [Derived] Grant SJ, Beauchamp MR, Blanchard CM, Carson V, Rhodes RE. Promoting sport participation during early parenthood: a randomized controlled trial protocol. Trials. 2020 Feb 27;21(1):230. doi: 10.1186/s13063-020-4158-x. PMID 32103772